CLINICAL TRIAL: NCT07182123
Title: The Influence of GLP1-RA on Periodontal Health - a Pilot Study
Brief Title: GLP1-RA and Periodontitis
Status: Not yet recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 1378/2025
Record Dates: First submitted 2025-09-11; First posted 2025-09-19 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Periodontitis; Diabetes (DM)
Keywords: periodontitis; diabetes; GLP1-RA
MeSH Terms: conditions — Periodontitis; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Periodontitis is among the most common chronic diseases worldwide and, along with caries, represents the leading cause of tooth loss. More recent theories regarding the etiology of periodontitis also attribute a significant role to the body's inflammatory response in the development and progression of the disease.

It is already well established that periodontitis is bidirectionally associated with other systemic inflammatory conditions, such as type 2 diabetes mellitus. Results from meta-analyses suggest that diabetes increases the likelihood of periodontal disease by approximately 24%, while periodontitis, conversely, raises the risk of type 2 diabetes by about 26%.

In addition to primary preventive measures and the modification of modifiable risk factors, diabetes mellitus is also treated pharmacologically with GLP-1 receptor agonists (GLP-1RA). In this context, Zhang et al. demonstrated that the administration of GLP-1RA, both in vitro and in vivo in rat models, leads to a significant reduction of pro-inflammatory substances in blood and periodontal tissue. However, to date, no clinical studies have investigated the effect of GLP-1RA on periodontal disease in humans.

For this reason, the aim of this pilot study is to investigate the effect of GLP-1RA on the periodontal status of patients with periodontitis. The data from this pilot study will subsequently be used to perform a power analysis to determine the sample size for a double-blind, placebo-controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent for participation and data protection
* Diagnosis of type 2 diabetes
* Diagnosis of chronic periodontitis (Caton, Armitage et al. 2018), presence of a PSI ≥ 3 in at least one sextant (Ainamo, Barmes et al. 1982)

Exclusion Criteria:

* Use of systemic antibiotics within the past 6 months
* Systematic periodontal treatment within the past 24 months
* Consumption of ≥ 5 cigarettes/day
* Unstable cardiovascular disease
* Chronic systemic diseases (e.g., rheumatoid arthritis, Crohn's disease, etc.)
* Pregnancy
* Use of the following medications: Immunosuppressants, Anticonvulsants, Calcium channel blockers
* Drug or medication abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be recruited during routine care at the Clinical Division of Endocrinology and Diabetology, University Hospital Graz, where treatment is provided in accordance with current clinical guidelines. In line with the S2k guideline "Interrelationships between Periodontal Diseases and Diabetes Mellitus", patients receive standardized education on the bidirectional association between periodontitis and diabetes, as this relationship is regarded as clinically relevant. As part of recommended care, an annual periodontal examination is scheduled; accordingly, patients are referred from endocrinological diagnostics to the Clinical Division of Conservative Dentistry, Periodontology, and Prosthodontics for baseline periodontal assessment (Sanz, Ceriello et al. 2018).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-10-24 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Effect of weekly GLP1-RA administration on periodontal clinical parameters (PD, CAL, BOP, furcation involvement, and tooth mobility) measured using a periodontal probe in patients with stage III or IV periodontitis. | From enrollment to the end of treatment at 16 weeks